CLINICAL TRIAL: NCT03568214
Title: Is Personalized Moderate Intensity Exercise Training Combined With High Intensity Interval Training More Effective at Improving Training Responsiveness When Compared to Moderate Intensity Exercise Training Alone?
Brief Title: Personalized Moderate Intensity Exercise Training Combined With High Intensity Interval
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Colorado University (Other)
Collaborators: Flinders University (Other)
Responsible Party: Principal Investigator, Lance Dalleck, Associate Professor, Western Colorado University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WesternSCU(3)
Record Dates: First submitted 2018-05-30; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Exercise; Metabolic Syndrome
Keywords: Primary Prevention
MeSH Terms: conditions — Motor Activity; Metabolic Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individualized moderate + high-intensity (Experimental): * 12 weeks of moderate-intensity continuous training (MICT) combined with high-intensity interval training (HIIT)
  * 4 days per week of MICT for 50 minutes per session
  * 1 day per week of HIIT for 35 minutes per session
  * Exercise intensity for MICT will be established according to ventilatory thresholds one and two (VT1 and VT2)
  * The HIIT protocol will consist of eight, 60 second intervals at 100% maximal oxygen uptake (VO2max), separated by 150 seconds active recovery
  Interventions: Other: Exercise
- Standardized moderate-intensity (Experimental): * 12 weeks of MICT
  * 5 days per week of MICT for 50 minutes per session
  * Exercise intensity for MICT will be established according to 40-65% heart rate reserve (HRR)
  Interventions: Other: Exercise
- Control (No Intervention): non-exercise control group testing at baseline and post-program (12 weeks)

INTERVENTIONS:
Other: Exercise — The MICT will be prescribed according to two exercise intensity methods: individualized (i.e., VT1 and VT2) and standardized (i.e., HRR). The HIIT will be prescribed based on individual fitness (i.e., VO2max).
  Arms: Individualized moderate + high-intensity; Standardized moderate-intensity

SUMMARY:
The purpose of this study will be to determine if personalized moderate intensity exercise training combined with high intensity interval training is more effective at improving training responsiveness than moderate intensity exercise training alone? This question will be addressed holistically be creating a composite score to assess training responsiveness. Additionally, individualized biological variability will be calculated in order to quantify training responsiveness using a personalized criterion. It is hypothesized that personalized moderate intensity exercise training combined with high intensity interval training will be more effective at improving comprehensive training responsiveness when compared to moderate intensity exercise training alone?

DETAILED DESCRIPTION:
It is well established that regular physical activity and cardiorespiratory fitness (CRF) training confers numerous health benefits and that a low level of CRF is a risk factor for coronary heart disease and cardiovascular disease (CVD) mortality. It is generally accepted that CRF can be improved with the implementation of a regular aerobic exercise training program following standardized guidelines. However, it has also been shown that not all individuals respond positively to such exercise, indeed there is considerable individual variability in training adaptations including so-termed 'non-responders' and, in some instances, 'adverse responders'. This variability in training responsiveness is not well understood and may be attributable to various factors including absence of a set definition in the literature for incidence of response and lack of an individualized approach to the exercise prescription.

It has been purported that a more individualized approach to the exercise prescription may enhance training efficacy and limit training unresponsiveness. For instance, it has been acknowledged as far back as the late 1970s that utilizing a relative percent method (i.e., % heart rate reserve [HRR]) to establish exercise intensity fails to account for individual metabolic responses to exercise. Nevertheless, the relative percent concept remains the gold standard recommendation for exercise intensity. It is both plausible and practical to think that an intensity set based on an individual's threshold measurement (i.e. ventilatory threshold) will not only encourage more positive physiological adaptations, but may account for some of the variability in training responsiveness by taking into consideration individual metabolic differences.

Additionally, high intensity interval training (HIIT) has emerged as a potential time efficient strategy for health promotion. Current recommended guidelines of 150 minutes of moderate physical activity per week is reduced by half to 75 minutes if the week's activity is done at a vigorous intensity. It has been demonstrated that HIIT, when compared to moderate intensity continuous training (MICT), has resulted in equal or superior improvements in VO2max, insulin action and sensitivity, endothelial function, systolic blood pressure, hip and waist circumference and lipid oxidation. The American College of Sports Medicine suggests considering incorporating interval training after a period of initial conditioning (typically 2-3 months) intermittently to avoid excessive orthopedic stress. Additionally, HIIT may require initial supervision in untrained and high risk individuals, and may transiently increase the risk of cardiac events in people with underlying undiagnosed CVD. Therefore, it seems pragmatic and consistent with current recommendations to combine the two types of training to achieve the greatest positive changes in cardiovascular and metabolic health.

It has been common practice to quantify training responsiveness based on absolute changes, but this method fails to take into consideration biological variability (normal day-to-day biological fluctuations) and measurement error of the equipment. Consequently, currently there is not a clear consensus on best practice to prescribe a customized exercise intervention that takes into consideration individual characteristics and diagnostic information. Furthermore, it may be that a personalized definition of biological variability is warranted. This is congruent with the line of reasoning that a more individualized approach to the exercise prescription may enhance training efficacy and limit training unresponsiveness. Simply put - if we are looking at exercise prescription (i.e., the front end) from an individualized perspective, it would also make sense to look at training responsiveness (i.e., the back end) from an individualized perspective as well.

Furthermore, classification and interpretation of training responsiveness may require a holistic view that integrates all exercise training outcomes. For example, in a recent study an adverse response in one single measure rarely resulted in higher overall risk of CVD. In fact, 10-year CVD risk increased in only three individuals (out of 332 individuals) as highlighted in this investigation. This finding has practical implications suggesting that although some individuals may have adverse or nonresponse cardiometabolic responses to exercise training, this may not always result in increased CVD risk and exercise may benefit these participants in different ways, such as improved cardiorespiratory fitness. Indeed, in the previously mentioned study, more than 40% (9/22) of 'adverse responders' concurrently increased cardiorespiratory fitness levels by 10% or more. Higher levels of cardiorespiratory fitness have been offered as an antidote toward other risk factors. Moreover, the literature suggests a 15% reduction in mortality for a 10% improvement in cardiorespiratory fitness. Taken together, it may be unintentionally misleading to categorize someone as an "adverse responder or non-responder to exercise" based on a single cardiometabolic factor when it is well known that regular exercise training confers a myriad of benefits. Clearly, the overall topic of training responsiveness to exercise warrants much additional study.

45 low-to-moderate risk, sedentary men and women will be recruited and randomized to one of the following arms:

* MICT + HIIT exercise program (N = 15)
* MICT exercise program (N = 15)
* non-exercise control group (N = 15)

ELIGIBILITY:
Inclusion Criteria:

* Considered low to moderate risk for cardiovascular disease based on the American College of Sports medicine guidelines
* Currently sedentary (participating in less than 30 minutes of moderate intensity physical activity on at least three days a week)
* Resided at an altitude of 2300 meters for at least the last 6 months

Exclusion Criteria:

* Any known sign, symptom, or diagnosed cardiovascular, pulmonary, metabolic, or similar disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2max) | 12 weeks
  gas exchange data measured with indirect calorimetry

SECONDARY OUTCOMES:
blood pressure | 12 weeks
  measured using a sphygmomanometer
fasting blood lipids and glucose | 12 weeks
  measured by analysis of a fingerstick blood sample using the Cholestech LDX System
waist circumference | 12 weeks
  measured using a cloth tape with a spring-loaded handle
body composition | 12 weeks
  measured via skinfold assessment
weight | 12 weeks
  measured with medical grade scale

CONTACTS AND LOCATIONS:
Overall Officials: Lance Dalleck, PhD, Principal Investigator — A/Professor and Institutional Officer
Locations (1):
- Western State Colorado University, Gunnison, Colorado, United States

IPD SHARING:
Plan to Share IPD: No